CLINICAL TRIAL: NCT02291081
Title: A Prospective, Epidemiologic and Multicentre Trial to Determine the Cardiovascular Risk, New Cardiovascular Events and the Cardiovascular Diseases in HIV-infected Patients: 10 Year Follow-up
Brief Title: A Prospective Observational Trial to Determine Cardiovascular Diseases in HIV-infected Patients
Acronym: HIV-HEART10
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Collaborators: Nico Reinsch M. D. (Unknown); Till Neumann Prof. M. D. (Unknown)
Responsible Party: Principal Investigator, Stefan Esser M.D., Academic director, University Hospital, Essen
Other Study IDs: 12-4970-BO A
Record Dates: First submitted 2014-10-21; First posted 2014-11-14 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: HIV-infection; Coronary Heart Disease; Myocardial Infarction; HIV-encephalopathy; Heart Failure; Aging
Keywords: HIV, AIDS; antiretroviral therapy; aging; heart failure; coronary heart disease; myocardial infarction; HIV-associated neurocognitive disorders
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Coronary Disease; Myocardial Infarction; AIDS Dementia Complex; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stored blood samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Comprehensive non invasive cardiovascular examination — Comprehensive non invasive cardiovascular examination
  * Anamnesis with the participants
  * File recherche,Physical examination
  * Documentation of the cardiovascular and antiretroviral medical therapy
  * Electrocardiogram
  * Transthoracic echocardiography
  * Exercise electrocardiogram
  * Exercise Montreal Cognitive Assessment test
  * Exercise the Grooved Pegboard test
  * Blood collection
  * Questionnaire to quality of life and health economics

SUMMARY:
The HIV/HEART study (HIVH) is an ongoing, prospective, multicentre trial that was conducted to assess the incidence, the prevalence and the clinical course of cardiovascular diseases (CVD) in HIV-infected patients. The study population includes outpatients from specialized HIV-care units of the German Ruhr region, who were at least 18 years of age, were known to have a HIV-infection and exhibited a stable disease status within 4 weeks before inclusion into the trial. From March 2004 (Pilot phase) to May 2014 (7,5 year Follow-up) 1481 HIV+ patients were recruited in a consecutive manner. The standardised examinations included a targeted assessment of medical history and physical examination. Blood was drawn for comprehensive laboratory tests including HIV specific parameters (CD4 cell count, HIV-1 RNA levels) and cardiovascular items (lipid concentrations, BNP values and renal parameters). Furthermore, non-invasive tests were performed during the initial visit, including additional heart rate and blood pressure measurements, electrocardiogram (ECGs) and transthoracic echocardiography (TTE). Examinations were completed in accordance with previously defined standard operating procedures. CVD were defined as coronary, cerebrovascular, peripheral arterial disease, heart failure or cardiac vitium.

DETAILED DESCRIPTION:
A comprehensive detailed description of the study procedures had been previously published (European Journal of medical research 2007;12:243-248).

Comprehensive non invasive cardiovascular examination

* Anamnesis
* File recherche,Physical examination
* Documentation of the cardiovascular and antiretroviral medical therapy
* Electrocardiogram
* Transthoracic echocardiography
* Exercise electrocardiogram
* Exercise Montreal Cognitive Assessment test
* Exercise the Grooved Pegboard test
* Blood collection
* Questionnaire to quality of life and health economics

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Known HIV-infection
* Written informed consent

Exclusion Criteria:

* Acute cardiovascular disease
* Unstable hemodynamic status in the three weeks before inclusion
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participiants were included in several cities of the Ruhrarea. Locations were Essen, Bochum, Dortmund and Duisburg The study population included outpatients who were at least 18 years of age, had a known HIV-infection and exhibited a stable disease status within 4 weeks before inclusion of the trial. Written informed consent was obtained from all participants.
Sampling Method: Non-Probability Sample
Enrollment: 1519 (Actual)
Dates: Start 2014-10; Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Diseases an deaths in HIV-infected Patients | Baseline up to 10 year follow-up

SECONDARY OUTCOMES:
Impact of classic cardiovascular risk factors and new HIV-specific risk factors of coronary artery disease, comorbidities and antiretroviral therapy | Baseline up to 10 year follow-up
  Patients included in the pilot-baseline trial and additionally in the 5 and 7.5 year follow-up will be recruited again for the 10 year follow-up after giving informed consent. After including a total of 1481 patients in the previous phases, now both therapy-naive patients as well as patients being treated with new agents should be included.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Esser, MD, Principal Investigator — Depatment of dermatology and venerology
Locations (7):
- Germany (7):
  - University Hospital of Bochum, Department of Dermatology, Bochum, North Rhine-Westphalia
  - City Hospital Dortmund, Dortmund, North Rhine-Westphalia
  - HIV physician pratice, Duisburg, North Rhine-Westphalia
  - University Hospital, Department of Dermatology and Venerology, Essen, North Rhine-Westphalia
  - HIV physician practice, Essen, North Rhine-Westphalia
  - HIV physician practice, Krefeld, North Rhine-Westphalia
  - Clinical Coordinating Center Leipzig, Leipzig, Saxony

REFERENCES:
- [Result] Neumann T, Woiwod T, Neumann A, Miller M, Von Birgelen C, Volbracht L, Esser S, Brockmeyer N, Gerken G, Erbel R. Cardiovascular risk factors and probability for cardiovascular events in HIV-infected patients - part III: age differences. Eur J Med Res. 2004 May 28;9(5):267-72. PMID 15257881
- [Result] Breuckmann F, Nassenstein K, Kondratieva J, Esser S, Erbel R, Potthoff A, Brockmeyer NH, Neumann T, Barkhausen J; German Heart Failure Network; Competence Network HIV/AIDS. MR characterization of cardiac abnormalities in HIV+ individuals with increased BNP levels. Eur J Med Res. 2007 May 29;12(5):185-90. PMID 17513188
- [Result] Neumann T, Esser S, Potthoff A, Pankuweit S, Neumann A, Breuckmann F, Neuhaus K, Kondratieva J, Buck T, Muller-Tasch T, Wachter R, Prettin C, Gelbrich G, Herzog W, Pieske B, Rauchhaus M, Loffler M, Maisch B, Mugge A, Wasem J, Gerken G, Brockmeyer NH, Erbel R; HIV-HEART Study Investigative Group. Prevalence and natural history of heart failure in outpatient HIV-infected subjects: rationale and design of the HIV-HEART study. Eur J Med Res. 2007 Jun 27;12(6):243-8. PMID 17666313
- [Result] Potthoff A, Brockmeyer NH, Gelbrich G, Neuhaus K, Esser S, Reinsch N, Hower M, Mostardt S, Neumann A, Neumann T; Competence Center Cardiac Insufficiency and the Competence Network HIV/AIDS. Lipodystrophy - a sign for metabolic syndrome in patients of the HIV-HEART study. J Dtsch Dermatol Ges. 2010 Feb;8(2):92-8. doi: 10.1111/j.1610-0387.2009.07330.x. Epub 2009 Dec 14. English, German. PMID 20002869
- [Result] Neumann T, Reinsch N, Neuhaus K, Brockmeyer N, Potthoff A, Esser S, Hower M, Neumann A, Mostardt S, Gelbrich G, Erbel R; fur die HIV-HEART-Studie sowie die Kompetenznetze Herzinsuffizienz und HIV/AIDS. [BNP in HIV-infected patients]. Herz. 2009 Dec;34(8):634-40. doi: 10.1007/s00059-009-3313-7. German. PMID 20024643
- [Result] Reinsch N, Neuhaus K, Esser S, Potthoff A, Hower M, Brockmeyer NH, Erbel R, Neumann T; German Competence Network for Heart Failure; German Competence Network for HIV AIDS. Prevalence of cardiac diastolic dysfunction in HIV-infected patients: results of the HIV-HEART study. HIV Clin Trials. 2010 May-Jun;11(3):156-62. doi: 10.1310/hct1103-156. PMID 20739268
- [Result] Reinsch N, Neuhaus K, Esser S, Potthoff A, Hower M, Mostardt S, Neumann A, Brockmeyer NH, Gelbrich G, Erbel R, Neumann T; German Competence Network Heart Failure; German Competence Network for HIV/AIDS. Are HIV patients undertreated? Cardiovascular risk factors in HIV: results of the HIV-HEART study. Eur J Prev Cardiol. 2012 Apr;19(2):267-74. doi: 10.1177/1741826711398431. Epub 2011 Feb 28. PMID 21450595
- [Result] Gelbrich B, Neumann T, Esser S, Potthoff A, Reinsch N, Hower M, Dannhauer KH, Loeffler M, Brockmeyer NH, Erbel R, Gelbrich G; HIV-HEART Study Investigative Group, Competence Networks Heart Failure and HIV/AIDS. Oral health and the heart - does HIV infection open a pathophysiological gateway? Int J Cardiol. 2011 Sep 1;151(2):254-7. doi: 10.1016/j.ijcard.2011.06.081. Epub 2011 Jul 18. No abstract available. PMID 21764468
- [Result] Esser S, Gelbrich G, Brockmeyer N, Goehler A, Schadendorf D, Erbel R, Neumann T, Reinsch N. Prevalence of cardiovascular diseases in HIV-infected outpatients: results from a prospective, multicenter cohort study. Clin Res Cardiol. 2013 Mar;102(3):203-13. doi: 10.1007/s00392-012-0519-0. Epub 2012 Nov 2. PMID 23117698
- [Result] Lind A, Reinsch N, Neuhaus K, Esser S, Brockmeyer NH, Potthoff A, Pankuweit S, Erbel R, Maisch B, Neumann T. Pericardial effusion of HIV-infected patients ? Results of a prospective multicenter cohort study in the era of antiretroviral therapy. Eur J Med Res. 2011 Nov 10;16(11):480-3. doi: 10.1186/2047-783x-16-11-480. PMID 22027640
- [Result] Reinsch N, Kahlert P, Esser S, Sundermeyer A, Neuhaus K, Brockmeyer N, Potthoff A, Erbel R, Buck T, Neumann T. Echocardiographic findings and abnormalities in HIV-infected patients: results from a large, prospective, multicenter HIV-heart study. Am J Cardiovasc Dis. 2011;1(2):176-84. Epub 2011 Jul 30. PMID 22254197